CLINICAL TRIAL: NCT07320066
Title: Reflections of Inspiratory Muscle Training on Patient Experiences in Asthma Rehabilitation
Brief Title: IMT in Asthma: Activity, Coping, Self-Management
Acronym: IMT in Asthma
Status: Recruiting | Type: Observational
Sponsor: Istanbul Esenyurt University (Other)
Responsible Party: Principal Investigator, Cahidenur Koçak, Principal investigator, Saglik Bilimleri Universitesi
Other Study IDs: IMT_Asthma_1
Record Dates: First submitted 2025-12-09; First posted 2026-01-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Qualitative Research
Keywords: asthma; inspiratory muscle training; telerehabilitation; self-management; qualitative research
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Rehabilitation Group (PRGr): Pulmonary Rehabilitation Group (PRGr)
  Participant selection for the study was conducted using a purposive sampling approach. All participants experienced inspiratory muscle training for a total of 3 days per week over 8 weeks, with 2 days per week via video conference and 1 day per week as part of a home program. All interviews will be conducted online via a video conference website and recorded using a digital voice recorder. The recorded data will be transcribed word for word in Turkish.
  Interventions: Other: other

INTERVENTIONS:
Other: other — Other: Telephone concept elicitation interview
  All interview questions are designed to be quite open-ended in order to determine participants' preferences in an unbiased manner (as much as possible). Additional questions will only be used when necessary to ensure that all relevant concepts are covered. Participants will be asked questions about the effects of inspirational muscle training they have previously experienced on their daily lives, coping strategies, and self-management processes.

SUMMARY:
The aim of this study is to investigate asthma patients' experiences with an 8 week IMT and the perceived effects of this intervention on physical activity, coping strategies, and asthma self-management. A qualitative methodological design will be applied to understand the experiences of patients participating in the IMT program, how the program affected their daily activities, how they coped with symptoms and difficulties, and how they managed their condition.

DETAILED DESCRIPTION:
The study will include patients diagnosed with asthma by a chest disease specialist and referred for pulmonary rehabilitation. Cases meeting the inclusion criteria will be questioned about the effects of their previous experience with COPD on their daily lives, their coping strategies, and their self-management processes. Therefore, it is determined as a basic criterion that participants have received IMT training for 8 weeks, 2 days a week via video conference and 1 day within the home program, for a total of 3 days a week. IMT should be performed in 7 sets, consisting of 2 minutes of work and 1 minute of rest, for a total of 21 minutes. Five main themes were identified as a result of data analysis. (a) Inspiratory Muscle Training and Participant Experiences (b) Experience of Exercising with Telerehabilitation (c) Changes in Physical Activity Levels (d) Self-Management Skills and (e) Coping Strategies.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having been diagnosed with severe persistent, non-allergic asthma by a pulmonologist in accordance with the Global Initiative for Asthma (GINA) guideline criteria,
* Patients with type 2 inflammation markers. According to accepted standards; peripheral eosinophils <150/µL and/or negative skin prick test and/or total IgE <30 kU/L
* Bronchodilator response (>12% or 200 mL improvement in FEV1% predicted following inhalation of 400 mg salbutamol)
* Diagnosis-follow-up period: Patients diagnosed at least 6 months prior, under follow-up and treatment, and/or with controlled asthma
* Having completed the pulmonary rehabilitation program
* Completion of 8 weeks of inspiratory muscle training (IMT)
* Patients who have read, understood, and signed the informed consent form

Exclusion Criteria:

* Having recently had a respiratory tract infection recently (within the last month),
* Having a smoking history of more than 10 pack-years or having a history of smoking within 6 months after quitting smoking
* Having received oral corticosteroid treatment in the last 4 weeks,
* Having a Body Mass Index >35,
* Eosinophilic Granulomatosis Polyangiitis (EGPA) and Allergic Bronchopulmonary Aspergillosis (ABPA),
* Vasculitis,
* History of malignancy,
* Pregnancy,
* Previous lung surgery, use of long-term oxygen therapy
* Having accompanying restrictive lung diseases (advanced kyphoscoliosis, ankylosing spondylitis) and neuromuscular diseases (myastania gravis, muscular dystrophies, myopathies) that will prevent healthy respiratory function testing and rehabilitation.
* Cognitive dysfunction, mental retardation, dementia, or other conditions that make it difficult to follow the protocol,
* Unwillingness to continue participating in the study,
* Communication difficulties or intellectual deficiencies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-19 (Estimated)

PRIMARY OUTCOMES:
Patient-reported experiences of inspiratory muscle training (IMT) assessed by semi-structured in-depth interviews (study-specific interview guide) | Single assessment after completion of the 8-week IMT program (within 4 weeks after IMT completion)
  Semi-structured, in-depth, audio-recorded interviews will be conducted using a study-specific interview guide containing open-ended questions to investigate the effect of an 8-week inspiratory muscle training (IMT) program on the experiences of adults with severe persistent asthma. Interviews will be conducted online and, when possible, in person or via telephone/video call. Interviews are expected to last approximately 45-60 minutes. Recordings will be transcribed verbatim in Turkish, supplemented with the researcher's field notes, and analyzed using thematic analysis.
Experience of exercising using telerehabilitation assessed by semi-structured in-depth interviews (study-specific interview guide) | Single assessment after completion of the 8-week IMT program (within 4 weeks after IMT completion)
  Semi-structured, in-depth, audio-recorded interviews will be conducted using a study-specific interview guide with open-ended questions to explore participants' experiences of exercising with telerehabilitation, including the perceived role of telerehabilitation in the learning process, and perceived advantages, limitations, and challenges from the participant's perspective. Interviews will be conducted online and, when possible, in person or via telephone/video call. Interviews are expected to last approximately 45-60 minutes. Recordings will be transcribed verbatim in Turkish, supplemented with the researcher's field notes, and analyzed using thematic analysis.
Changes in physical activity in daily life assessed by semi-structured in-depth interviews (study-specific interview guide) | Single assessment after completion of the 8-week IMT program (within 4 weeks after IMT completion)
  Semi-structured, in-depth, audio-recorded interviews will be conducted using a study-specific interview guide with open-ended questions to explore perceived changes in physical activity in daily life (e.g., walking, climbing stairs, housework) from the participant's perspective following the 8-week program. Interviews will be conducted online and, when possible, in person or via telephone/video call. Interviews are expected to last approximately 45-60 minutes. Recordings will be transcribed verbatim in Turkish, supplemented with the researcher's field notes, and analyzed using thematic analysis.
Self-management skills assessed by semi-structured in-depth interviews (study-specific interview guide) | Single assessment after completion of the 8-week IMT program (within 4 weeks after IMT completion)
  Semi-structured, in-depth, audio-recorded interviews will be conducted using a study-specific interview guide with open-ended questions to explore participants' perceived self-management skills, including disease and trigger recognition, symptom monitoring, accountability/responsibility, and perceived control. Interviews will be conducted online and, when possible, in person or via telephone/video call. Interviews are expected to last approximately 45-60 minutes. Recordings will be transcribed verbatim in Turkish, supplemented with the researcher's field notes, and analyzed using thematic analysis.
Coping strategies assessed by semi-structured in-depth interviews (study-specific interview guide) | Single assessment after completion of the 8-week IMT program (within 4 weeks after IMT completion)
  Semi-structured, in-depth, audio-recorded interviews will be conducted using a study-specific interview guide with open-ended questions to explore participants' perceived coping strategies, including breathing/respiratory rate control strategies and emotional and behavioral regulation during symptom attacks and when anxiety/panic symptoms are prominent. Interviews will be conducted online and, when possible, in person or via telephone/video call. Interviews are expected to last approximately 45-60 minutes. Recordings will be transcribed verbatim in Turkish, supplemented with the researcher's field notes, and analyzed using thematic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Esenyurt University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided